CLINICAL TRIAL: NCT06743243
Title: Effect of Tegoprazan for Elective Surgery Patients Under General Anesthesia
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Seok Kyeong Oh (Other)
Collaborators: Korea University Guro Hospital (Other); HK inno.N Corporation (Industry); Eunpyeong St. Mary's Hospital, The Catholic University of Korea (Unknown); Asan Medical Center (Other)
Responsible Party: Sponsor-Investigator, Seok Kyeong Oh, Professor of Anesthesiology, Korea University Guro Hospital
Organization: Korea University Guro Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KCAB_032
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: General Anesthesia
Keywords: K-CAB; K-CAB OD tab.; P-CAB; Famotidine; Tegoprazan; general anesthesia
MeSH Terms: interventions — tegoprazan; Famotidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group T (Experimental): Tegoprazan OD tab. 50 mg PO + Saline 20 ml IV, one hour before general anesthesia.
  Interventions: Drug: Tegoprazan
- Group F (Active Comparator): Famotidine 20 mg/10 ml + Saline 10 ml IV + Tegoprazan OD tab. 50 mg placebo PO, one hour before general anesthesia.
  Interventions: Drug: Famotidine
- Group C (Placebo Comparator): Tegoprazan OD tab. 50 mg placebo PO + Saline 20 ml IV, one hour before general anesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan OD tab. 50 mg PO + Saline 20ml IV, one hour before general anesthesia.
  Arms: Group T
Drug: Famotidine — Famotidine 20mg/10ml+saline 10ml IV + Tegoprazan OD tab. 50 mg placebo PO, one hour before general anesthesia.
  Arms: Group F
Drug: Placebo — Tegoprazan OD tab. 50 mg placebo PO + Saline 20ml IV, one hour before general anesthesia.
  Arms: Group C

SUMMARY:
The aim of this study is to compare gastric pH right after endotracheal intubation for general anesthesia in patients pretreated with tegoprazan, famotidine, or placebo.

DETAILED DESCRIPTION:
This clinical trial is a prospective, randomized, double-blind, multicenter, investigator-initiated trial that aims to demonstrate the preventive effect of tegoprazan on preoperative aspiration in patients scheduled to undergo surgery using general anesthesia.

Subjects who meet the inclusion/exclusion criteria will be randomly assigned to the tegoprazan administration group (Group T), famotidine administration group (Group F), or placebo administration group (Group C) in the same ratio of 1:1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Has a plan to undergo surgery with general anesthesia with inhalation or total Intravenous
2. Subjects aged between 20 and 69 years
3. ASA classification I - III

Exclusion Criteria:

1. Conduct Emergency surgery
2. BMI(Body Mass Index) ≥ 35
3. Has a history of drug abuse or depandency.
4. Has a history of Anesthetic allergy
5. Has a plan to undergo resection(gastric cancer, esophageal cancer)

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Gastric pH right after endotracheal intubation | right after endotracheal intubation

SECONDARY OUTCOMES:
Change of oral, esophageal and gastric pH | oral pH(before anesthesia, endotracheal intubation 30 minutes after surgery started, right after surgery end, extubation, 30minutes after enter the postanesthesia care unit), esophageal and gastric pH(right after intubation)
Gastric volume evaluated by Ultrasound | before anesthesia, right after end of surgery, 30 minutes after enter the postanesthesia care unit
Risk of aspiration(pH < 2.5, Gastric volume > 0.4mL/kg) and frequency of complications(aspiration etc.) | before anesthesia, right after intubation, 30 minutes after surgery started, right after surgery end, extubation, 30 minutes after enter the postanesthesia care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Medical Center, Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided